CLINICAL TRIAL: NCT05359809
Title: The Effect of Grasping Palmar Reflex on Pain and Stress in Peripheral Intravenous Central Catheter Intervention in Preterm Infants
Brief Title: Peripheral Intravenous Central Catheter Intervention in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Collaborators: MSc İknur Budancamanak (Unknown)
Responsible Party: Principal Investigator, Türkan Kadiroğlu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.O.01.00/264
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Preterm; Pain, Acute; Stress; Nursing Caries
Keywords: Preterm; Pain, Acute; Stress; Nursing Caries
MeSH Terms: conditions — Premature Birth; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grasping Palmar Reflex (Experimental)
  Interventions: Behavioral: Graspin Palmar Reflex Stimulation
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Graspin Palmar Reflex Stimulation — The grasping reflex is an involuntary response involving the hands and fingers. flexion-adduction movement. The reflex resembles the grasping movement of the hand. The reflex can be achieved by moving an object distally across the palm.
  Arms: Grasping Palmar Reflex

SUMMARY:
This study will be conducted to evaluate the effect of grasping reflex stimulation applied during peripheral intravenous central catheter (PIC) intervention on pain and stress in preterm infants receiving treatment and care in the neonatal intensive care unit.

DETAILED DESCRIPTION:
The study was planned in a parallel randomized controlled trial design. The population of the research will be preterm infants followed in the Newborn Intensive Care Unit of Atatürk University Health Research and Application Center between May 2022 and September 2022. Randomization in the sample of the study will be done in the computer environment. Sample size was determined by power analysis. In the collection of data; Preterm Baby Information Form, Preterm Baby Follow-up Form, Neonatal Stress Scale and ALPS-NEO pain and stress assessment scale will be used. In the control group, the PIC intervention will be performed by the investigator in accordance with clinical procedures. In the experimental group, the baby's grasping reflex stimulation will be provided during the PIC attempt.

ELIGIBILITY:
Inclusion Criteria:

* Between 26-32 weeks of gestation,
* Birth weight of 1500 g and below,
* No congenital defects
* who need PIC intervention while receiving treatment and care in the NICU,
* Not receiving sedation at least 3 hours before the PIC procedure,
* No neurological problems
* No surgical intervention
* Recipient of noninvasive mechanical ventilation
* infants whose parents approved the informed voluntary consent form

Exclusion Criteria:

* Painful procedure (invasive procedure, etc.) has been performed in the last hour,
* Infants without parental informed consent form

Ages: 26 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Pain Level | 12 week
  Neonatal pain and stress rating scale: The scale was developed by Lundqvist et al. in 2014. It is used to measure pain and stress in preterm and term newborns. The scale is a five-item scale that includes the newborn's facial expression, breathing pattern, tone of the extremities, hand and foot activity, and activity level. The lowest score that can be obtained from the scale is 0 and the highest score is 10. As the scale score increases, it indicates that the level of pain and stress increases.
Stress Levell | 12 week
  Neonatal stress scale: It was developed to evaluate stress in premature babies. The scale consists of eight items; facial expression, body color, respiration, activity level, comfortability, muscle tone, extremities, and posture. Scale It is a 3-point Likert type and is evaluated between 0-2 points in scoring. A minimum of 0 points from the scale, A maximum of 16 points is taken. As the score increases, the baby's stress level increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No